CLINICAL TRIAL: NCT01668498
Title: Comparison of Two Preemptive Treatment Strategies of Panitumumab Mediated Skin Toxicity and Assessment of Quality of Life in Patients With Ras-wildtype Colorectal Cancer
Brief Title: Comparison of Two Preemptive Treatment Strategies of Panitumumab Mediated Skin Toxicity and Assessment of QoL in Patient With Ras-wt Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AIO-LQ-0110; 2010-022938-85 (EudraCT Number)
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Ras-wildtype Colorectal Cancer
Keywords: Can preemptive treatment of panitumumab mediated skin; toxicity with oral doxycycline be replaced by local treatment with erythromycin?; Panitumumab
MeSH Terms: interventions — Erythromycin; erythromycin, ammonium bituminosulfonate drug combination; Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erythromycin (Experimental): Experimental Arm (ARM A) skin- treatment: erythromycin cream 2% daily at bedtime doxycycline 100mg b.i.d.if skin toxicity CTC° ≥2 skin moisturizer daily at morning, sunscreen before going outdoors for 8 weeks
  Interventions: Drug: Erythromycin
- Doxycyline (Active Comparator): Standard Arm (ARM B) skin- treatment:doxycycline 100mg b.i.d. skin moisturizer daily at morning, sunscreen before going outdoors for 8 weeks
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Erythromycin — Comparison of efficacy of Arm A erythromycin cream 2% daily at bedtime (doxycycline 100mg b.i.d.if skin toxicity CTC° ≥2) and Arm B doxycycline 100mg b.i.d. in patients with Metastatic Colorectal cancer (Ras wild-type)being treated with panitumumab.
  Other Names: Aknemycin
  Arms: Erythromycin
Drug: Doxycycline — Comparison of efficacy of Arm A erythromycin cream 2% daily at bedtime (doxycycline 100mg b.i.d.if skin toxicity CTC° ≥2) and Arm B doxycycline 100mg b.i.d. in patients with Metastatic Colorectal cancer (Ras wild-type)being treated with panitumumab.
  Arms: Doxycyline

SUMMARY:
80 - 90 % of the patients treated with anti-EGFR antibodies (panitumumab or cetuximab) experience skin toxicity, mostly acne like skin rash.

A standardized treatment of skin rash is neither established as standard arm for clinical trials nor as guideline for the treatment of skin toxicity in clinical practice. While an improvement of QoL has been demonstrated for panitumumab and cetuximab in comparison to best supportive care the data basis for patient related outcomes regarding skin toxicity deriving from randomized trials is still small.

Recent surveys among German oncologist revealed that physicians are reluctant to use oral antibiotics as preemptive treatment . Only 19 out of 110 oncologists stated that they are thinking about using preemptive treatment in patients with acne-like skin rash.

Thus, in the present trial two main questions will be addressed:

(i) Can preemptive treatment with oral doxycycline be replaced by a sequential skin treatment strategy (i.e. local treatment with erythromycin followed by doxycycline in case of inefficacy = development of acne) without compromising treatment efficacy of skin toxicity treatment? (ii) Comparison of general and skin related QoL between both treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with wild-type RAS (KRAS and NRAS) status of metastatic colorectal cancer treatment with panitumumab according to label

   * RAS wild-type tested in
   * KRAS exon 2 (codons 12/13)
   * KRAS exon 3 (codons 59/61)
   * KRAS exon 4 (codons 117/146)
   * NRAS exon 2 (codons 12/13)
   * NRAS exon 3 (codons 59/61)
   * NRAS exon 4 (codons 117/146)
2. treatment with pre-emptive study medication shall begin the day before treatment start with panitumumab
3. Willingness to cope with biweekly quality of life questionnaires
4. Written Informed consent
5. Aged at least 18 years
6. ECOG Performance Status 0-2
7. Life expectancy of at least 12 weeks
8. Adequate haematological, hepatic, renal and metabolic function parameters:

   * Leukocytes > 3000/mm³
   * ANC ≥ 1500/mm³
   * Platelets ≥ 100,000/mm³
   * Haemoglobin > 9 g/dl
   * Serum creatinine ≤ 1.5 x ULN
   * Bilirubin ≤ 1.5 x ULN
   * GOT-GPT ≤ 2.5 x ULN (in case of liver metastases GOT / GPT ≤ 5 x ULN)
   * AP ≤ 5 x ULN
   * Magnesium, Calcium and potassium within normal ranges (may be substituted before study entry)

Exclusion criteria:

1. Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment.
2. Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment (adequate: oral contraceptives, intrauterine device or barrier method in conjunction with spermicidal jelly).
3. Serious concurrent diseases
4. On-treatment participation in a clinical study in the period 30 days prior to inclusion
5. Clinically significant cardiovascular disease in (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrolment.
6. History of interstitial lung disease, e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.
7. History of HIV infection.
8. Other previous or concurrent malignancy (≤ 5 years prior to enrolment in study) except non-melanoma skin cancer or cervical carcinoma FIGO stage 0- 1 if the patient is continuously disease-free
9. Known allergic reactions on panitumumab, doxycycline or erythromycin
10. Previous treatment with anti-cancer agents directed against EGFR (e.g. cetuximab, panitumumab, erlotinib, gefitinib, lapatinib)
11. Skin rash existing before or due to other reasons than panitumumab treatment
12. Other dermatologic disease that may interfere with correct grading of panitumumab induced skin rash
13. Parallel treatment with anti-tumor agents other than panitumumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-05; Primary Completion 2015-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients developing no skin toxicity ≥ grade 2 | 8 weeks
  Percentage of patients developing no skin toxicity ≥ grade 2 at any time during their first 8-weeks of treatment with panitumumab.

SECONDARY OUTCOMES:
Quality of life | 8 weeks
  Quality of life will be assessed by standardized skin-related (DLQI) and global quality of life (EORTC QLQ C30.
  For correlation analyses between the different quality of life scores, the non-parametric test according to Spearman will preferably be applied.
Assess Skin toxicity | 8 weeks
  Assess different skin toxicity grading scales (i.e. NCI CTC v. 4.0; WoMo score; MESTT)
Correlation between skin-related and global quality of life | 8 weeks
  Description of correlation between skin-related and global quality of life using EORTC-QLQ C30 and SF-36.
late skin toxicity | from week 8 to 12
  Describe the development of late skin toxicity after 8 weeks
Skin-toxicity related dose reductions of panitumumab | 8 weeks
  Rate of skin-toxicity induced dose reductions (including withdrawal) of panitumumab

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Kripp, Dr. med., Principal Investigator — III. Medizinische Klinik, Universitätsmedizin Mannheim
Locations (1):
- Universitätsklinikum Mannheim, III. Medizinische Klinik, Mannheim, Germany

REFERENCES:
- See also: Related Info — http://www.aio-portal.de